CLINICAL TRIAL: NCT05971888
Title: Impact and Process Evaluation of the Better Dairy for All Program in Ethiopia
Brief Title: Better Dairy for All Evaluation in Ethiopia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The program, Better Dairy for All, funded by the Global Alliance for Improved Nutrition (GAIN) will no longer continue because of state of emergency imposed in Amhara Region, making it infeasible to implement programmatic activities.
Sponsor: RTI International (Other)
Collaborators: Bahir Dar University (Other); Frontieri Consult (Unknown)
Responsible Party: Principal Investigator, Valerie Flax, Senior Research Public Health Analyst, RTI International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 424603
Record Dates: First submitted 2023-07-20; First posted 2023-08-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Dairy Consumption
Keywords: diet; dairy; market intervention; social and behavior change communication intervention; children; workers; Ethiopia

STUDY DESIGN:
Intervention Model Description: Data will be collected through household surveys, worker surveys, dairy value chain actor surveys, in-depth interviews (IDIs), and focus group discussions (FGDs). In Amhara Region, the protocol team has selected a subset of the intervention districts for the evaluation and identified an equal number of districts outside the program coverage area with similar characteristics to serve as the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Food system and demand generation
- Control (No Intervention): In Amhara, an equal number of districts outside the program coverage area with characteristics similar to the intervention districts will serve as the control.

INTERVENTIONS:
Behavioral: Food system and demand generation — GAIN's program to increase dairy consumption among BoP children and workers will include components to increase demand, improve access, and support the enabling environment. In Amhara, the demand generation component will share messages through radio, community influencers, and community conversations led by health extension workers targeting rural BoP households with children 6 months up to 7 years. GAIN will train milk houses and cooperatives on dairy safety and quality assurance and better business practices and will assist with cold chain and milk dispensing technology to improve milk availability and access. In industries and large-scale farms, GAIN will use a demand generation strategy to inform workers about the importance of dairy products and other nutritious foods and to encourage them to purchase them at their workplaces. GAIN will work with local businesses to launch and maintain dairy dispensers and arrange provision of other nutritious foods at work sites.
  Arms: Intervention

SUMMARY:
Global Alliance for Improved Nutrition (GAIN)'s "Better Dairy for All" program in Ethiopia seeks to improve children's and workers' consumption of healthy foods by improving access, increasing demand, and improving the enabling environment for dairy products by operating at multiple levels - individuals, households, markets, producers, and policies. RTI and local partners propose to conduct impact and process evaluations of GAIN's program tailored to the theory of change. The evaluation will include a mix of quantitative and qualitative methods and will be guided by the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) evaluation framework.

DETAILED DESCRIPTION:
Background: Dairy products are excellent sources of calcium, vitamin A, and vitamin B12, and good sources of zinc, but are not widely consumed in Ethiopia. GAIN's Better Dairy for All program has two main components. One component is focused on increasing dairy consumption among children 6 months up to 7 years in bottom of the pyramid (BoP) households in Amhara Region through a demand generation campaign and support to milk houses, cooperatives, and processors. The other component is focused on increasing consumption of dairy and other nutritious foods by BoP workers in industries and large-scale farms by making dairy and other nutritious foods, such as fortified oil and fortified wheat flour and fruits/vegetables, available at their workplaces accompanied by demand generation activities.

Objective: The objective of this study is to conduct an impact and process evaluation of GAIN's Better Dairy for All program.

Methods: In Amhara, the evaluation will use a parallel group mixed-methods quasi-experimental before-after design to assess the effectiveness of the intervention on dairy consumption of children. The evaluation will be carried out in 64 enumeration areas (EAs) in intervention woredas matched on demographic characteristics with 64 EAs in control woredas. Data will be collected through household surveys, semi-structured interviews with dairy value chain actors, and focus group discussions (FGDs) with caregivers of young children. Cross-sectional population-based household surveys with caregivers of young children will be conducted at baseline (N=1,144) and endline (N=1,144) to assess intervention impact on dairy consumption frequency and quantity using difference-in-differences analysis. In the intervention woredas, evaluators will conduct semi-structured interviews to evaluate program outcomes with milk houses, milk processors, and cooperatives (N=30) at baseline, midline, and endline. Evaluators will also conduct FGDs with caregivers of young children (N=8 FGDs) at midline and endline in the intervention woredas. This data will be used for the process evaluation.

In industries and large-scale farms, the evaluation of GAIN's program will use a cross-sectional pre-post design. The evaluation will be carried out in 5 purposefully selected industries/farms that start the intervention around the same time. Data will be collected through worker surveys, in-depth interviews (IDIs), and FGDs. Surveys with workers (N=524) will be conducted before and after the intervention to measure impacts of the program on workers' dairy consumption frequency and quantity. IDIs with industry/farm owners or managers and suppliers of dairy and other nutritious foods (N=5-10) and IDIs with workers (N=15) will be conducted at midline and endline. This data will be used for process evaluation.

ELIGIBILITY:
Household surveys

Inclusion Criteria:

* Reside in the enumeration areas;
* Be a caregiver of at least one child 6 months to 7 years old residing in the enumeration area;
* Be over 18 years old;
* The household is classified as BoP on Poverty Probability Index;
* Be able to speak Amharic;
* Provide informed consent to participate in the study.

Dairy value chain semi-structured interviews

Inclusion Criteria:

* Be a manager or owner of small and medium enterprises (milk houses, milk processors, or cooperatives) in the districts selected for the evaluation;
* Be over 18 years old;
* Be able to speak Amharic;
* Provide informed consent to participate in the study.

FGDs with caregivers

Inclusion criteria:

* Be a caregiver of a child 6 months up to 7 years old living in the intervention districts selected for the evaluation;
* Be over 18 years old;
* Be able to speak Amharic;
* Provide informed consent to participate in the study.

Worker surveys

Inclusion criteria:

* Be a worker at an industry or large-scale farm where the owner/manager has agreed to participate in GAIN's program;
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Amharic;
* Provide informed consent to participate in the study.

In-depth interviews with workers

Inclusion criteria:

* Be an owner, worker, or food supplier connected to industries or large-scale farms involved in GAIN's program in the intervention districts selected for the evaluation;
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Amharic;
* Provide informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of dairy consumption | Baseline (August 2023), Endline (July 2026) (3 years)
  Description (limit 999 characters) Change in the mean frequency of dairy consumption during the last 7 days by children 6 months to 7 years and workers
Frequency of nutritious food consumption | Baseline (August 2023), Endline (July 2026) (3 years)
  Change in the mean frequency of consumption of promoted nutritious foods (fortified oil, wheat flour, and fruits/vegetables) during the last 7 days by workers

SECONDARY OUTCOMES:
Number of available dairy and nutritious foods | Baseline (August 2023), Endline (July 2026) (3 years)
  Change in number of available dairy and target nutritious foods

CONTACTS AND LOCATIONS:
Overall Officials: Netsanet Fentahun, PhD, Principal Investigator — Bahir Dar University
Locations (1):
- Frontieri, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be shared through Nesstar.